CLINICAL TRIAL: NCT03102047
Title: A Phase II Study to Assess the Activity of PD-L1 Inhibition With Durvalumab (MEDI4736) After Chemo-Radiotherapy in Patients With Stage II-IV Microsatellite Stable (MSS) Rectal Cancer
Brief Title: Study of Durvalumab (MEDI4736) After Chemo-Radiation for Microsatellite Stable Stage II-IV Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FR-2; ESR-15-11477 (Other: AstraZeneca)
Record Dates: First submitted 2017-03-07; First posted 2017-04-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Rectal Cancer
Keywords: microsatellite stable; MSS; durvalumab; NSABP
MeSH Terms: conditions — Rectal Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- durvalumab (Experimental): IV infusion once every 2 weeks for 4 total doses
  Interventions: Drug: durvalumab

INTERVENTIONS:
Drug: durvalumab — Within 3-7 days after completion of chemoradiation, patients will receive durvalumab (750 mg IV infusion) every 2 weeks for 4 doses on Day 1(Dose 1), Day 15 (Dose 2), Day 29 (Dose 3), and Day 43 (Dose 4)
  Other Names: MEDI4736

SUMMARY:
This study is being done to look at the safety and response to the investigational drug durvalumab (MEDI4736) following chemo-radiation therapy for patients with MSS stage II to IV rectal cancer. Durvalumab recognizes specific proteins on the surface of cancer cells and triggers the immune system to destroy the cancer cells. The chemoRT portion of the treatment will be completed just before the course of durvalumab is initiated.

In order to learn more about certain characteristics of rectal cancer tumors, this study includes special research tests using samples from diagnostic tumors, a tissue sample from tumors removed during surgery, fresh tumor samples from an area where the cancer has recurred, and blood samples.

DETAILED DESCRIPTION:
The FR-2 study is designed as a phase II, open label, single arm study in patients with microsatellite stable (MSS) stages II-IV rectal cancer, to assess the activity of PD-L1 inhibition with durvalumab (MEDI4736) monotherapy after standard chemo-radiotherapy (chemoRT). The study's primary aim is to determine the safety and efficacy of durvalumab immediately following chemoRT in patients undergoing subsequent surgery with stage II-IV rectal cancer.

One dose of durvalumab will be given every 2 weeks for four total doses beginning within 3-7 days of completing chemoRT. Surgery for all patients must occur within 8-12 weeks of the final dose of RT. Adjuvant chemotherapy after surgical recovery is at the discretion of the treating physician.

During a safety run-in, the first 6 patients will be closely followed for 30 days after last dose of durvalumab without further accrual of patients. Patients will receive durvalumab (750mg IV infusion once every 2 weeks) for 4 total doses. No other concurrent anti-neoplastic medications or treatments aside from standard supportive care will be allowed during the durvalumab treatment phase.

The safety run-in portion of the study will proceed to full enrollment at the proposed study therapy dose, (750 mg IV infusion every 2 weeks), if one or less dose-limiting toxicity (DLT) or significant safety concern attributable to durvalumab is identified during the observation period of the first 6 patients. If there are two or more DLTs, accrual to the study will stop with reassessment of the protocol.

A total of 44 patients will be enrolled in this study for a sample size of 41 surgically evaluable patients.

Required tissue and blood samples will be collected at specific time points and submitted for correlative science studies. Optional tumor and blood samples will be collected from consenting patients upon disease recurrence or progression.

Given the increasing use of non-operative therapy for patients with rectal cancer who achieve a complete clinical response and in order to maximize the inclusion of patients participating in this trial, the primary endpoint was changed from NAR score to modified NAR score (mNAR). The mNAR score substitutes values from clinical staging for the pathologic T-Stage and N-Stage for those patients who don't go to surgery because of a complete clinical response and consequently have no pathology. Additionally, because of enrollment challenges related to COVID-19 pandemic and the exploratory nature of including stage IV patients, the stage IV analysis was moved to exploratory and reducing the number of patients needing to be enrolled in the study to approximately 44.

ELIGIBILITY:
Inclusion Criteria:

* The ECOG performance status must be 0 or 1
* Patients with biopsy-proven adenocarcinoma, stage II- IV rectal cancer.
* The tumor must have been determined to be mismatch repair proficient or microsatellite stable through CLIA approved testing (Immunohistochemistry [IHC], polymerase chain reaction [PCR], or Next-Generation Sequencing [NGS] assays).
* Patients must be candidates for planned surgical resection of their primary rectal cancer 8 - 12 weeks after completion of neoadjuvant chemoRT, even if stage IV.
* Planned neoadjuvant chemoRT treatment must conform to NCCN guidelines.
* Baseline staging prior to chemoRT initiation must be obtained. If stage IV, there must be documentation by PET/CT scan, CT scan, or MRI, that the patient has evidence of measurable distant disease per RECIST 1.1. Note: Patients with stage IV disease should have limited but measurable metastatic disease (one or two organs involved e.g., liver and lung) and primary tumor deemed resectable.
* Blood counts performed within 4 weeks prior to study entry must meet the following criteria:

  * ANC must be greater than or equal to 1500/mm3
  * Platelet count must be greater than or equal to 75,000/mm3; and
  * Hemoglobin must be greater than or equal to 9 g/dL.
* Adequate hepatic function performed within 4 weeks prior to study entry must be met:

  * Total bilirubin must be less than or equal to 1.5 x ULN (upper limit of normal) for the lab unless the patient has a bilirubin elevation greater than 1.5 x Upper limit of normal (ULN) to 3 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
  * AST and ALT must be less than or equal to 2.5 x ULN for the lab with the following exception: for patients with documented liver metastases, AST and ALT must be less than or equal to 5 x ULN.
* Adequate renal function within 4 weeks of study entry, defined as serum creatinine less than or equal to 1.5 x ULN for the lab. (If creatinine is 1.0-1.5 x ULN, the creatinine clearance should be greater than 40 mL/min per Cockcroft-Gault formula (Cockcroft-Gault 1976), or by 24-hour urine collection for determination of creatinine clearance.)
* Patients with reproductive potential (male/female) must agree to use accepted and highly effective methods of contraception while receiving durvalumab, and for at least 3 months after the last dose of durvalumab.

Exclusion Criteria:

* Diagnosis of anal or small bowel carcinoma.
* Histopathology other than adenocarcinoma, e.g., sarcoma, lymphoma, carcinoid.
* Previous therapy with any PD1 or PD-L1 inhibitor (including durvalumab) for any malignancy.
* Completion of pelvic radiotherapy treatment for this current rectal cancer or any prior pelvic radiotherapy (e.g., prior prostate or cervical cancer therapy).
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days after receiving the last dose of durvalumab.
* Acute or chronic hepatitis B or hepatitis C.
* Known history of human immunodeficiency virus (HIV) or acquired immunodeficiency-related (AIDS) illnesses.
* History of brain metastases, uncontrolled spinal cord compression, carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
* Active infection or chronic infection requiring chronic suppressive antibiotics.
* History of allogeneic organ transplantation.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* Active or prior history of autoimmune or inflammatory condition requiring ongoing immunosuppressive medications. This specifically includes use of immunosuppressive medication within 28 days before the first dose of durvalumab with the exceptions of intranasal corticosteroids or systemic corticosteroids at physiological doses, which do not exceed 10mg/day of prednisone or an equivalent corticosteroid.
* Any of the following cardiac conditions:

  * Documented NYHA Class III or IV congestive heart failure
  * Myocardial infarction within 6 months prior to study entry
  * Unstable angina within 6 months prior to study entry
  * Symptomatic arrhythmia
* Uncontrolled high blood pressure defined as systolic BP greater than or equal to 150 mmHg or diastolic BP greater than or equal to 100 mmHg with or without anti-hypertensive medication. Patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria.
* Ongoing or active gastritis or peptic ulcer disease.
* Active bleeding diatheses which in the opinion of the treating physician poses a significantly increased operative risk.
* Known history of previous diagnosis of tuberculosis.
* History of hypersensitivity to durvalumab or any excipient.
* Known history of active pneumonia, pneumonitis, symptomatic interstitial lung disease, or definitive evidence of interstitial lung disease described on CT scan, MRI, or chest x-ray in asymptomatic patients; dyspnea at rest requiring current continuous oxygen therapy.
* Other malignancies unless the patient is considered to be disease-free and has completed therapy for the malignancy greater than or equal to 12 months prior to study entry. Patients with the following cancers are eligible if diagnosed and treated within the past 12 months: carcinoma in situ of the cervix, colorectal carcinoma in situ, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements, or interfere with interpretation of study results.
* Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing should be performed within 14 days prior to study entry according to institutional standards for women of childbearing potential.)
* Use of any investigational agent within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Median modified Neoadjuvant Rectal (mNAR) Score | From the beginning of the study to time of surgical resection, assessed over an estimated 12 weeks
  Compare Median modified Neoadjuvant Rectal (mNAR) Score to historic control using the Wilcoxon test

SECONDARY OUTCOMES:
Pathologic complete response rate to study therapy | At the time of surgical resection
  Pathologic Complete response rate ( pCR) (ypT0 and ypN0) of primary rectal cancer and regional nodes determined by pathological examination
Clinical complete response rate to study therapy | From one week prior to surgical resection up to time of surgical resection
  Clinical complete response rate cCR (ycT0) determined by the clinical absence of the primary tumor via digital rectal exam and proctoscopic exam
Rate of negative circumferential margin | At the time of surgical resection
  Rate of negative circumferential margin in surgical resection specimens
Sphincter function in patients with sphincter preserving surgery | From the time of surgical resection to 30 days after surgery
  Sphincter function as determined by number of adverse events related to bowel control
Severity of post-operative complications | From time of surgical resection to within 30 days post-operation
  Surgical complications that result in re-hospitalizations or death
Frequency of adverse events assessed by CTCAE 4.0 | From beginning of study therapy to 90 days after last dose of study therapy
  Frequency of adverse events categorized using the NCI Common Terminology Criteria for Adverse Events version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (43):
- United States (43):
  - Smilow Cancer Hospital Care Center at Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Yale, New Haven, Connecticut
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center at North Haven, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital at Lawrence + Memorial Cancer Center, Waterford, Connecticut
  - University of Florida, Gainesville, Florida
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Cancer Care Specialists of Central Illinois-Crossroads Cancer Center, Effingham, Illinois
  - Cancer Care Specialists of Central Illinois-Swansea, Swansea, Illinois
  - University of Michigan Oncology, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Strecker Cancer Center, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Columbus NCORP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates, Inc., Delaware, Ohio
  - Delaware Health Center Grady Cancer Center, Delaware, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Marion General Hospital, Marion, Ohio
  - The Mark H. Sangmeister Center, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Port Clinton, Ohio
  - Genesis Health Care Center, Zanesville, Ohio
  - UPMC Hillman Cancer at Upper St Clair, Bethel Park, Pennsylvania
  - UPMC Hillman Cancer Center at Mt. View, Greensburg, Pennsylvania
  - AHN Cancer Institute at Jefferson, Jefferson Hills, Pennsylvania
  - Forbes Regional Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center at Monroeville, Monroeville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - WPAON/Medical Center Clinic, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital dba West Penn Hospital, Pittsburgh, Pennsylvania
  - UPCI Hillman/Shadyside, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at Passavant OHA, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center at Passvant HOA, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center at Washington, Washington, Pennsylvania
  - West Virginia University Medicine, Morgantown, West Virginia
  - West Virginia University, Morgantown, West Virginia